CLINICAL TRIAL: NCT01227772
Title: A Phase I/IIa Study of OTSGC-A24 Vaccine in Advanced Gastric Cancer
Brief Title: Study of OTSGC-A24 Vaccine in Advanced Gastric Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Wakayama Medical University (Other); Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA04/26/10
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer vaccine; OTSGC-A24; A Phase I/IIa study; HLA-A24-positive
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weekly Cohort (Experimental): The gastric cancer vaccine (OTSGC-A24) will be administered at a dose of 1 mg once a week
  Interventions: Biological: OTSGC-A24
- 2-weekly cohort (Experimental): The gastric cancer vaccine (OTSGC-A24) will be administered at the dose of 1 mg every 2 weeks.
  Interventions: Biological: OTSGC-A24
- 3-weekly cohort (Experimental): The gastric cancer vaccine (OTSGC-A24)will be administered at 1 mg very 3 weeks
  Interventions: Biological: OTSGC-A24

INTERVENTIONS:
Biological: OTSGC-A24 — OTSGC-A24 administered at 1 mg in weekly, 2-weekly, and 3-weekly cohorts.

SUMMARY:
Active vaccination with tumor specific antigens and VEGFR1 HLA-A24 epitopes can improve survival of patients with advanced Gastric Cancer.

DETAILED DESCRIPTION:
Although palliative chemotherapy improved the outcome of patients with advanced Gastric Cancer, the prognosis for this group of patients remains poor. Tumor specific antigens and angiogenesis pathway are potential targets for immunotherapy. A cocktail of peptide vaccines is selected to overcome gastric cancer's heterogeneous and enhance the anti-tumor effect. Five HLA-A*2402-binding peptide vaccines derived from tumor specific antigens and VEGFR1 are chosen based on the frequencies of their expressions in gastric cancer and the ability to induce specific cytotoxic T-lymphocytes. In preclinical model, both down regulation these targets with siRNA and active vaccination resulted in tumor regression. The purpose of the study is to evaluate the safety and optimal dosing schedule of a cancer vaccine cocktail, OTSGC-A24 targeting novel specific tumor antigens FOXM1, DEPDC1, KIF20A, URLC10 and VEGFR1 in advanced gastric cancer patients with HLA-2402 haplotype.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed inoperable or metastatic adenocarcinoma of the stomach or lower third of the oesophagus refractory or intolerable to standard therapy.
* Patients must have measurable or evaluable disease.
* Age >= 201years
* ECOG performance status of 0 to 2
* Life expectancy at least 3 months
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count >=1,500/mcL
* platelets >=100,000/mcL
* total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) <=2.5 X institutional upper limit of
* Normal creatinine within normal institutional limits
* Patients must be HLA-A*2402
* Patients must have recover from all reversible treatment toxicity from prior chemotherapy, radiotherapy or surgery.
* The effects of OTSGC-A24 on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients receiving any other investigational agents.
* History of significant gastrointestinal bleeding that required intervention within the prior 1 month is ineligible; inherited bleeding diathesis or coagulopathy.
* Serious non healing wound and peptic ulcer disease
* Previous history of intestinal perforation
* Invasive procedures defined as follows (Insertion of a vascular access device is not considered major/minor surgery):
* Major surgical procedure, open biopsy or significant traumatic injury =28 days prior to -registration
* Anticipation of need for major surgical procedures during the course of the study
* Core biopsy <=7 days
* Minor surgery <=2 weeks
* Symptomatic CNS metastasis
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, uncontrolled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg), symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction/cerebrovascular event (<=6 months prior to study entry), cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, long term systemic immunosuppressant or corticosteroid.
* Women who are breast-feeding or pregnant are excluded from this study

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
safety of OTSGC-24 | within 4 weeks of treatment
  Dose limiting toxicity will be evaluated during the first 4 weeks of treatment. If in the unlikely event that DLT is observed in 1 of the 3 subjects, an additional 3 subjects will be enrolled at the same dose level. If DLT is observed in 2 of the 6 subjects, subsequent cohorts will be treated at 0.5 mg.
Optimal dosing schedule | 1 year
  In each cohort, OTSGC-A24 (~1 mg) will be administered subcutaneously at 3-weekly (cohort 1), 2-weekly (cohort 2) and weekly (cohort 3) interval. Treatment may continue until the subject experiences confirmed disease progression or unacceptable toxicity, withdraws consent, or requires treatment with another therapeutic modality.

SECONDARY OUTCOMES:
Induction of specific cytotoxic T-lymphocyte (CTL) response | after 4 weeks and 12 weeks of vaccination
  Up to 10 patients per cohort will be recruited in the cohort or cohorts with the highest specific CTL induction rate to define the optimal dosing schedule for OTSGC-A24.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Peng Yong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Wakayama Medical University Hospital, Wakayama, Japan
- National University Hospital, Singapore, Singapore, Singapore
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Background] Ajani JA. Evolving chemotherapy for advanced gastric cancer. Oncologist. 2005;10 Suppl 3:49-58. doi: 10.1634/theoncologist.10-90003-49. PMID 16368871
- [Background] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Derived] Sundar R, Rha SY, Yamaue H, Katsuda M, Kono K, Kim HS, Kim C, Mimura K, Kua LF, Yong WP. A phase I/Ib study of OTSGC-A24 combined peptide vaccine in advanced gastric cancer. BMC Cancer. 2018 Mar 27;18(1):332. doi: 10.1186/s12885-018-4234-8. PMID 29587677